CLINICAL TRIAL: NCT02045238
Title: Study of the Effect of Inhaled 3% Hypertonic Saline Compared With Normal Saline (0,9%) for the Treatment of Acute Viral Bronchiolitis in a Short Stay Ward
Brief Title: Inhaled Hypertonic Saline Use in the Emergency Department to Treat Acute Viral Bronchiolitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulties (reduced staff plus university strike)
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mateus Deckers Leme, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1263/13 - University Hospital
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Therapeutics; Saline Solution, Hypertonic
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic; X-Rays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): Patients will receive inhaled normal saline, initially with a 2 hour interval, and clinical evaluation prior to each inhalation. When they attain sat>94% AND respiratory rate <60 AND RDAI score <4, the interval between inhalations will be changed to 4 hours. If they maintain these criteria for a whole 4 hour interval, they are discharged. If they do not improve enough to be discharged in 24 hours from the first inhalation, they are considered as admitted to hospital.
  Interventions: Radiation: Chest X-Ray; Other: Respiratory virus screening test
- Hypertonic Saline (Experimental): Patients will receive inhaled Hypertonic Saline 3%, initially with a 2 hour interval, and clinical evaluation prior to each inhalation. When they attain sat>94% AND respiratory rate <60 AND RDAI score <4, the interval between inhalations will be changed to 4 hours. If they maintain these criteria for a whole 4 hour interval, they are discharged. If they do not improve enough to be discharged in 24 hours from the first inhalation, they are considered as admitted to hospital.
  Interventions: Drug: Hypertonic Saline; Radiation: Chest X-Ray; Other: Respiratory virus screening test

INTERVENTIONS:
Drug: Hypertonic Saline — Sodium Chloride 3% solution, previously prepared in 5 mL syringes.
  Arms: Hypertonic Saline
Radiation: Chest X-Ray
Other: Respiratory virus screening test — Immunofluorescence analysis of nasal aspirate

SUMMARY:
Acute viral bronchiolitis is an extremely common childhood disease, responsible for approximately 17% of childhood admissions to hospital per year, with an annually cost that reaches U$ 500 million.

Despite being a well known disease among pediatricians, there are few, if any, effective treatment options apart from oxygen supplementation and adequate hydration.

The purpose of this study is to determine wether nebulized hypertonic saline (3%) is more effective than normal saline (0,9%) when used in repeated doses during the first 24 hours of in-hospital treatment.

DETAILED DESCRIPTION:
Acute viral bronchiolitis is a lower airway infection, caused manly by Respiratory Syncytial Virus. Near 1% of children up to 2 years of age get it with sufficient severity to warrant hospital admission, with an annual cost of about U$ 500 million in the US, superior, for instance, than cystic fibrosis annual cost.

Despite the physiopathology and clinical course being well known among pediatricians, few therapeutical options other than adequate hydration and oxygen supplementation have proven to be effective Corticosteroids are not effective and bronchodilators are controversial, and treatment is still mostly empiric and lacking evidence.

In the last few years, there has been a growing interest in the use of nebulized hypertonic saline (HS) as a promising approach. The rational is that HS would help reducing edema and mucus viscosity, enhancing its rheologic properties. Recent studies suggest that HS could reduce up to 1 day (25%) of time until discharge in admitted patients. In the Emergency Department, HS was not superior to other forms of treatment, but these studies lack power and similarities to draw further conclusions. Also, time of treatment and ideal interval between doses are not known as yet.

To our knowledge, few if any studies have assessed patients with an intermediary (up to 24h) time of stay, namely a short stay ward attached to an emergency department. Thus, we have endeavoured to determine if repeated doses of nebulized HS are superior to nebulized normal saline (NS) during the first 24 hour of treatment, when considered: rate of admission, time until discharge, time until attain discharge criteria, and rate of readmission after discharge.

Furthermore, most studies use HS associated to a bronchodilator, because of a theoretical possibility that HS alone could induce bronchoconstriction and worsen respiratory symptoms. However, recent studies have shown that HS use without bronchodilators have not caused any worsening of symptoms in bronchiolitis patients. Therefore, we propose to study the effect of HS alone, without the adding of bronchodilators, which would minimize bias in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Age < 12 months
* Clinical diagnosis of bronchiolitis (viral respiratory disease and wheezing)
* First episode of wheezing in life
* Moderate respiratory distress, defined as 2 of the following: Sat <93%, respiratory rate >60 and/or RDAI score >4

Exclusion Criteria:

* Previous episodes of wheezing in history
* Use of bronchodilators, corticosteroids or antibiotics in the 24 hours prior to admission or at any time during treatment.
* Other clinical conditions such as: prematurity, bronchopulmonary dysplasia, cystic fibrosis, cardiac disease or immunodeficiencies.
* detection of alveolar infiltrates suggestive of pneumonia in radiologic examination
* respiratory impairment requiring mechanical ventilation on arrival to hospital.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mateus D Leme, MD, Principal Investigator — Sao Paulo University
Locations (1):
- University Hospital of Sao Paulo University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Anil AB, Anil M, Saglam AB, Cetin N, Bal A, Aksu N. High volume normal saline alone is as effective as nebulized salbutamol-normal saline, epinephrine-normal saline, and 3% saline in mild bronchiolitis. Pediatr Pulmonol. 2010 Jan;45(1):41-7. doi: 10.1002/ppul.21108. PMID 19953579
- [Background] Mandelberg A, Tal G, Witzling M, Someck E, Houri S, Balin A, Priel IE. Nebulized 3% hypertonic saline solution treatment in hospitalized infants with viral bronchiolitis. Chest. 2003 Feb;123(2):481-7. doi: 10.1378/chest.123.2.481. PMID 12576370
- [Background] Kuzik BA, Al-Qadhi SA, Kent S, Flavin MP, Hopman W, Hotte S, Gander S. Nebulized hypertonic saline in the treatment of viral bronchiolitis in infants. J Pediatr. 2007 Sep;151(3):266-70, 270.e1. doi: 10.1016/j.jpeds.2007.04.010. Epub 2007 Jun 29. PMID 17719935
- [Background] Zhang L, Mendoza-Sassi RA, Wainwright C, Klassen TP. Nebulised hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2013 Jul 31;(7):CD006458. doi: 10.1002/14651858.CD006458.pub3. PMID 23900970
- [Background] Principi T, Komar L. A critical review of "a randomized trial of nebulized 3% hypertonic saline with epinephrine in the treatment of acute bronchiolitis in the emergency department.". J Popul Ther Clin Pharmacol. 2011;18(2):e273-4. Epub 2011 May 16. No abstract available. PMID 21633141
- [Background] Jacobs JD, Foster M, Wan J, Pershad J. 7% Hypertonic saline in acute bronchiolitis: a randomized controlled trial. Pediatrics. 2014 Jan;133(1):e8-13. doi: 10.1542/peds.2013-1646. Epub 2013 Dec 16. PMID 24344111
- [Background] Mandelberg A, Amirav I. Hypertonic saline or high volume normal saline for viral bronchiolitis: mechanisms and rationale. Pediatr Pulmonol. 2010 Jan;45(1):36-40. doi: 10.1002/ppul.21185. No abstract available. PMID 20014350
- [Background] Kuzik BA, Flavin MP, Kent S, Zielinski D, Kwan CW, Adeleye A, Vegsund BC, Rossi C. Effect of inhaled hypertonic saline on hospital admission rate in children with viral bronchiolitis: a randomized trial. CJEM. 2010 Nov;12(6):477-84. doi: 10.1017/s1481803500012690. PMID 21073773
- See also: University Hospital of Sao Paulo University — http://www.hu.usp.br

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline: Patients will receive inhaled normal saline, initially with a 2 hour interval, and clinical evaluation prior to each inhalation. When they attain sat>94% AND respiratory rate <60 AND RDAI score <4, the interval between inhalations will be changed to 4 hours. If they maintain these criteria for a whole 4 hour interval, they are discharged. If they do not improve enough to be discharged in 24 hours from the first inhalation, they are considered as admitted to hospital.
  Chest X-Ray
  Respiratory virus screening test: Immunofluorescence analysis of nasal aspirate
- Hypertonic Saline: Patients will receive inhaled Hypertonic Saline 3%, initially with a 2 hour interval, and clinical evaluation prior to each inhalation. When they attain sat>94% AND respiratory rate <60 AND RDAI score <4, the interval between inhalations will be changed to 4 hours. If they maintain these criteria for a whole 4 hour interval, they are discharged. If they do not improve enough to be discharged in 24 hours from the first inhalation, they are considered as admitted to hospital.
  Hypertonic Saline: Sodium Chloride 3% solution, previously prepared in 5 mL syringes.
  Chest X-Ray
  Respiratory virus screening test: Immunofluorescence analysis of nasal aspirate
Period: Overall Study
Arm/Group | Normal Saline | Hypertonic Saline
Started | 16 | 15
Completed | 9 | 14
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Population: Number of patients completing the study was too low to make statistically significant comparisons.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Hypertonic Saline | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  Brazil | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Rate of Admission
Description: Patients staying longer than 24h are considered to be admitted to ward.
Time Frame: 24 hours
Population: Number of participants analyzed was too small to obtain statistic significance
Measure: Number; unit: participants
Arm/Group | Normal Saline | Hypertonic Saline
Number analyzed (Participants) | 9 | 14
participants | 3 | 6

2. Primary Outcome: Time to Attain Discharge Criteria
Description: Discharge criteria are: Room air saturation >94% AND respiratory rate < 60 AND Respiratory Distress Assessment Instrument (RDAI) score inferior than 4, maintained over a 4 hour period.
Time Frame: 24 hours
Reporting Status: Not Posted

3. Secondary Outcome: Time to Discharge
Description: Actual time to discharge was considered of secondary importance as it can be influenced by individual considerations like patient age or time of the day.
Time Frame: 24 hours
Reporting Status: Not Posted

4. Secondary Outcome: Rate of Readmission After Discharge
Description: The mere attendance to the Emergency Department will not be isolately considered, as it may be due to a scheduled reevaluation.
Time Frame: 5 days
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Adverse Effects
Description: Any adverse effects directly attributable to treatment shall be noted. Mere lack of improve or worsening of symptoms attributable to the disease clinical course will not be considered as adverse effects.
Time Frame: 24 hours
Population: Number of patients too small to achieve statistical significance
Measure: Number; unit: participants
Arm/Group | Normal Saline | Hypertonic Saline
Number analyzed (Participants) | 9 | 14
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Normal Saline | Hypertonic Saline
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/9 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes